CLINICAL TRIAL: NCT00441116
Title: An Randomised, Double-blind, Placebo-controlled, Parallel Group Study to Assess the Efficacy and Safety of Dutasteride 0.5mg Once Daily for 6 Months in the Treatment of Male Subjects With Androgenetic Alopecia (Norwood-Hamilton Classification Type IIIv, IV and V)
Brief Title: A Study To Assess The Efficacy And Safety Of Dutasteride 0.5mg Once Daily For 6 Months In The Treatment Of Male Subjects With Androgenetic Alopecia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 106377
Record Dates: First submitted 2007-02-27; First posted 2007-02-28 (Estimated); Results first posted 2009-04-22 (Estimated); Last update posted 2018-08-16 (Actual); Status verified 2018-07

CONDITIONS: Alopecia
Keywords: dutasteride; Androgenic alopecia; phase 3
MeSH Terms: conditions — Alopecia | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- Dutasteride (Placebo Comparator): Dutasteride
  Interventions: Drug: Dutasteride 0.5mg oral tablets

INTERVENTIONS:
Drug: Dutasteride 0.5mg oral tablets — Dutasteride

SUMMARY:
The aim of this Phase III study is to compare the efficacy, safety and tolerability of dutasteride (0.5mg) with placebo for 6 months, in Korean male subjects with androgenetic alopecia in the vertex region, types IIIv, IV and V according to the modified Norwood-Hamilton Classification.

ELIGIBILITY:
Inclusion criteria:

* Rationale - The vertex area of the scalp will be evaluated during this study, therefore the inclusion criterion of Norwood Hamilton areas IIIv, IV or V ensures that subjects with vertex hair loss will be recruited in line with the primary efficacy endpoint of change in hair growth in the vertex.

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Male out-patients aged 18-49 years, inclusive
2. Diagnosis of Male Pattern Hair Loss classified as type IIIv, IV, or V utilising the modified Norwood-Hamilton classification (Figure 1) (N.B. types IVa and Va are excluded)
3. Able to comprehend instructions and record required information
4. Will provide signed and dated written informed consent to participate in this investigation

Exclusion criteria:

* A subject will not be eligible for inclusion in this study if any of the following criteria apply:

  1. Evidence of hypogonadism defined as serum testosterone < 250ng/dl and/or LH >20mIU/ml Note: If the initial serum testosterone result is < 250ng/dl and the LH value is normal, the test may be repeated once. Attempts should be made, where possible, to collect all samples in the morning hours. If the repeat testosterone result is < 250ng/dl, the subject is not eligible for participation.
  2. Greater than two times the upper limit of normal for ALT or AST, or a bilirubin greater than 2.0mg/dl (exception - subjects diagnosed with Gilbert's syndrome will be eligible to participate in the study)
  3. Serum creatinine >1.8mg/dl
  4. Global scalp hair thinning, including occipital areas
  5. Scarring of the scalp or any other condition or disease of the scalp or hair, including diseases of the hair shaft (e.g., uncontrolled seborrheic dermatitis, tinea infections, other causes of alopecia, prior hair transplants or scalp reductions, psoriatic dermatitis) and inability to discontinue use of hair weaving.
  6. Subjects who use hair colourants/hair dyes, or have the remaining traces of colourants in their hair. Subjects must maintain their natural hair colour throughout the study.
  7. Hair length in non-balding areas ≤2cm (3/4 inch) around the vertex region of the head. Subjects must maintain the same hairstyle throughout the study.
  8. History of malignancy within the past five years, except basal cell or squamous cell carcinoma of the skin
  9. Serum PSA level > 2.0 ng/ml at screening visit.
  10. Family history(Father, brothers) of prostate cancer.
  11. Active unstable thyroid disease, including subjects on therapy for either hyperthyroidism or hypothyroidism unless their dose of thyroid medication has been stable for 3 months and serum TSH is normal
  12. Hypersensitivity to any 5 AR inhibitor or drugs chemically related to the study medication
  13. Use of finasteride or other 5 AR inhibitors within the 12 months prior to screening.
  14. Previous use of dutasteride.
  15. Use of phytotherapy (e.g. saw palmetto) within 8 weeks prior to screening.
  16. Previous use of cytotoxic agents
  17. Use of glucocorticoids (inhaled glucocorticoids are allowed; topical steroids are allowed provided that they are not used on the scalp) within the 3 months prior to screening
  18. Use of the following during the 6 months prior to screening:

      * Minoxidil (oral or topical)
      * Drugs with anti-androgenic properties (e.g., cyproterone acetate, spironolactone, ketoconazole, flutamide, bicalutamide). Cimetidine cannot be used during the study but is not an excluded drug when used during the previous 6 months.
      * Topical estrogen, progesterone
      * Tamoxifen
      * Drugs potentially causing hypertrichosis (e.g., cyclosporine, diazoxide, phenytoin psoralens)
      * Anabolic steroids
      * Lithium and phenothiazines

  17. Concurrent or regular use during the 4 weeks prior to screening of topical agents to the scalp (e.g., anti-inflammatories) 18. Participation in any investigational or marketed drug trial within 30 days preceding the screening phase of this study. Participation in any other drug trial during the course of this study including the follow-up period.

  19. History or current evidence of drug or alcohol abuse within the 12 months prior screening 20. History of any illness (including psychiatric) which may impair the ability to provide informed consent or comply with study requirements 21. History of any unstable illness or condition that, in the opinion of the investigator, might confound the results or put the subject at risk.

  22. Subjects who are known to be HIV positive (status which includes subjects with AIDS) 23. Subjects who will not refrain from donating blood until completing the study follow-up period.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 153 (Actual)
Dates: Start 2006-12-15 (Actual); Primary Completion 2008-01-21 (Actual); Study Completion 2008-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Dutasteride: Subjects who were given 0.5mg of Dutasteride once daily for 6 months in male subjects age 18-49 years with Androgenetic Alopecia(AGA) in the vertex region, types IIIv, IV and V according to the modified Norwood-Hamilton Classification.
- Placebo: Subjects who were given no Investigational product.
Period: Overall Study
Arm/Group | Dutasteride | Placebo
Started | 76 | 77
Completed | 73 | 75
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Did not meet Eligibility Criteria | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dutasteride | Placebo | Total
Number analyzed (Participants) | 76 | 77 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.78 (7.07) | 38.41 (6.61) | 38.097 (6.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 76 | 77 | 153
Region of Enrollment [Number; unit: participants]
  Korea, Democratic People's Republic of | 76 | 77 | 153 (0) [0 to 0]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Hair Growth Assessed by Macrophotographic Technique (Hair Count) in the Vertex at 6 Months.
Description: The Macrophotographic hair count method marks a 1-inch diameter circular area at the anterior leading edge of the vertex thinning area and then photographed. The photographs are enlarged and converted into dot maps and the dot maps are converted into total hair counts by means of personal computer-based scanners and imaging software.
Time Frame: Baseline and 6 months
Population: Intent to Treat (ITT) population defined as all randomized subjects received at least one dose of study medication and having at least one on visit endpoint.
Measure: Mean (Standard Deviation); unit: hair count per centimeters squared
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
hair count per centimeters squared
  Baseline | 148.14 (36.27) | 144.27 (32.33)
  Month 6 | 162.27 (38.52) | 149.57 (34.44)
  Change from Baseline - Month 6 | 12.21 (23.60) | 4.67 (16.81)
Statistical Analysis 1: Comparison: Dutasteride vs Placebo; Month 6 - Baseline; Test type: Superiority or Other; p = 0.0319, t-test, 2 sided; Median Difference (Final Values) = 7.54, 95% CI [0.75 to 14.33], Standard Deviation 20.37 — Mean difference = Drug A minus Drug B

2. Secondary Outcome: Change From Baseline Hair Growth Assessed by Macrophotographic Technique (Hair Count) in the Vertex at 3 Months.
Description: as for outcome 1
Time Frame: Baseline and Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hair count per centimeters squared
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
hair count per centimeters squared
  Baseline | 148.14 (36.27) | 144.27 (32.33)
  Month 3 | 160.19 (36.73) | 154.50 (36.87)
  Change from Baseline - Month 3 | 7.58 (22.70) | 10.24 (19.02)

3. Secondary Outcome: Subjects Global Assessment of Hair Regrowth Question: Since the Start of Treatment I Have Lost?
Description: GlaxoSmithKline - Hair Growth Index without Photographs subject assessment of change in hair loss and overall appearance at 3 and 6 months. Subjects answered 4 questions without photographs concerning their perception of Change in Hair Growth.
Time Frame: Month 3 and Month 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Much less hair (Month 3) | 5 | 4
  Moderately less hair (Month 3) | 8 | 7
  Slightly less hair (Month 3) | 26 | 26
  The same amount of hair (Month 3) | 32 | 36
  Slightly more hair (Month 3) | 1 | 2
  Moderately more hair (Month 3) | 1 | 0
  Much more hair (Month 3) | 0 | 0
  Much less hair (Month 6) | 9 | 7
  Moderately less hair (Month 6) | 13 | 8
  Slightly less hair (Month 6) | 24 | 22
  The same amount of hair (Month 6) | 25 | 35
  Slightly more hair (Month 6) | 2 | 3
  Moderately more hair (Month 6) | 0 | 0
  Much more hair (Month 6) | 0 | 0

4. Secondary Outcome: Subjects Global Assessment of Hair Regrowth Question: Since the Start of Treatment my Usual Hair Loss Has Slowed Down?
Description: as for outcome 3
Time Frame: Month 3 and Month 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  I strongly disagree (month 3) | 0 | 1
  I disagree (month 3) | 18 | 30
  No opinion either way (month 3) | 20 | 13
  I agree (month 3) | 34 | 30
  I strongly agree (month 3) | 1 | 1
  I strongly disagree (month 6) | 0 | 0
  I disagree (month 6) | 18 | 27
  No opinion either way (month 6) | 12 | 17
  I agree (month 6) | 40 | 29
  I strongly agree (month 6) | 3 | 2

5. Secondary Outcome: Subjects Global Assessment of Hair Regrowth Question: Since Start of Treatment the Overall Appearance (Thickness, Hair Quality, Amount) of the Hair on my Head is?
Description: as for outcome 3
Time Frame: Month 3 and Month 6
Population: Intent to Treat (ITT) population defined as all randomized subjects received at least one dose of study mediction and having at least one on visit endpoint.
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Much worse (Month 3) | 0 | 0
  Moderately worse (Month 3) | 0 | 1
  Slightly worse (Month 3) | 1 | 4
  Not Changed (Month 3) | 36 | 47
  Slightly Better (Month 3) | 25 | 20
  Moderately Better (Month 3) | 7 | 3
  Much Better (Month 3) | 4 | 0
  Much worse (Month 6) | 0 | 0
  Moderately worse (Month 6) | 1 | 0
  Slightly worse (Month 6) | 2 | 10
  Not changed (Month 6) | 23 | 33
  Slightly Better (Month 6) | 26 | 29
  Moderately Better (Month 6) | 11 | 3
  Much Better (Month 6) | 10 | 0

6. Secondary Outcome: Subjects Global Assessment of Hair Regrowth Question: Since the Start of Treatment I Have Kept What Hair I Had?
Description: as for outcome 3
Time Frame: Month 3 and Month 6
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  I strongly disagree (Month 3) | 0 | 0
  I disagree (Month 3) | 4 | 8
  No opinion either way (Month 3) | 5 | 11
  I agree(Month 3) | 62 | 56
  I strongly agree (Month 3) | 2 | 0
  I strongly disagree (Month 6) | 0 | 0
  I disagree (Month 6) | 3 | 8
  No opinion either way (Month 6) | 3 | 9
  I agree (Month 6) | 60 | 58
  I strongly agree(Month 6) | 7 | 0

7. Secondary Outcome: Subjects Global Assessment of Hair Regrowth Question: Since the Start of Treatment, When I Look at my Thinning Area, I Can See?
Description: GlaxoSmithKline - Hair Growth Index with Photographs subject assessment of change in hair loss and overall appearance at 3 and 6 months. Subjects answered 4 questions comparing photographs of their hair before treatment and concerning the last week and evaluated the change in Hair Growth.
Time Frame: Month 3 and Month 6
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Much less scalp (month 3) | 10 | 3
  Moderately less scalp (month 3) | 17 | 11
  Slightly less scalp (month 3) | 25 | 17
  The same amount of scalp (month 3) | 14 | 26
  Slightly more scalp (month 3) | 3 | 14
  Moderately more scalp (month 3) | 1 | 4
  Much more scalp (month 3) | 3 | 0
  Much less scalp (month 6) | 9 | 2
  Moderately less scalp (month 6) | 16 | 5
  Slightly less scalp (month 6) | 26 | 15
  The same amount of scalp (month 6) | 20 | 26
  Slightly more scalp (month 6) | 1 | 22
  Moderately more scalp (month 6) | 1 | 4
  Much more scalp (month 6) | 0 | 1

8. Secondary Outcome: Subjects Global Assessment of Hair Regrowth Question: Since the Start of Treatment my Hair Now Covers?
Description: as for outcome 7
Time Frame: Month 3 and Month 6
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Much less scalp (Month 3) | 1 | 1
  Moderately less scalp (Month 3) | 2 | 3
  Slightly less scalp (Month 3) | 3 | 14
  The same amount of scalp (Month 3) | 20 | 24
  Slightly more scalp (Month 3) | 25 | 23
  Moderately more scalp (Month 3) | 15 | 7
  Much more scalp (Month 3) | 7 | 3
  Much less scalp (Month 6) | 0 | 2
  Moderately less scalp (Month 6) | 0 | 5
  Slightly less scalp (Month 6) | 2 | 21
  The same amount of scalp (Month 6) | 22 | 28
  Slightly more scalp (Month 6) | 17 | 17
  Moderately more scalp (Month 6) | 28 | 1
  Much more scalp (Month 6) | 4 | 1

9. Secondary Outcome: Subjects Global Assessment of Hair Regrowth Question: Since the Start of Treatment the Amount of Hair on my Thinning Area Has?
Description: as for outcome 7
Time Frame: Month 3 and Month 6
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Greatly decreased (Month 3) | 0 | 0
  Moderately decreased (Month 3) | 2 | 1
  Slightly decreased (Month 3) | 7 | 19
  Stayed the same (Month 3) | 17 | 21
  Slightly increased (Month 3) | 26 | 21
  Moderately increased (Month 3) | 15 | 10
  Greatly increased (Month 3) | 6 | 3
  Greatly decreased (Month 6) | 0 | 2
  Moderately decreased (Month 6) | 0 | 4
  Slightly decreased (Month 6) | 0 | 22
  Stayed the same (Month 6) | 22 | 26
  Slightly increased (Month 6) | 22 | 18
  Moderately increased (Month 6) | 23 | 2
  Greatly increased (Month 6) | 6 | 1

10. Secondary Outcome: Subjects Global Assessment of Hair Regrowth Question: Since the Start of Treatment the Appearance (Thickness, Hair Quality, Amount) of the Thinning Area on my Head is?
Description: as for outcome 7
Time Frame: Month 3 and Month 6
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Much Worse (Month 3) | 0 | 0
  Moderately Worse (Month 3) | 2 | 1
  Slightly Worse (Month 3) | 2 | 9
  Not Changed (Month 3) | 16 | 28
  Slightly Better (Month 3) | 28 | 24
  Moderately Better (Month 3) | 14 | 9
  Much Better (Month 3) | 11 | 4
  Much Worse (Month 6) | 0 | 1
  Moderately Worse (Month 6) | 0 | 2
  Slightly Worse (Month 6) | 0 | 20
  Not Changed (Month 6) | 21 | 25
  Slightly Better (Month 6) | 24 | 23
  Moderately Better (Month 6) | 19 | 2
  Much Better (Month 6) | 9 | 2

11. Secondary Outcome: Investigator's Photographic Assessment of Improvement Distribution From Baseline
Description: Improvement Distribution is based on the number of hairs per centimeters squared by macrophotographic conversion hair count. Score Range -3=greatly decreased to +3=greatly increased. 0=No change.
Time Frame: Month 3 and Month 6
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Greatly decreased (Month 3) | 0 | 0
  Moderately decreased (Month 3) | 1 | 1
  Slightly decreased (Month 3) | 0 | 13
  No Change (Month 3) | 28 | 30
  Slightly increased (Month 3) | 35 | 30
  Moderately increased (Month 3) | 8 | 1
  Greatly increased (Month 3) | 1 | 0
  Greatly decreased (Month 6) | 0 | 0
  Moderately decreased (Month 6) | 0 | 8
  Slightly decreased (Month 6) | 4 | 16
  No Change (Month 6) | 24 | 36
  Slightly increased (Month 6) | 31 | 14
  Moderately increased (Month 6) | 12 | 1
  Greatly increased (Month 6) | 2 | 0

12. Secondary Outcome: Investigator's Photographic Assessment of Improvements From Baseline Score
Description: Improvement Distribution Score is based on the number of hairs per centimeters squared by macrophotographic conversion hair count. Score Range: -3 = greatly decreased to +3 = greatly increased. 0 = No change.
Time Frame: Month 3 and Month 6
Population: Per Protocol Population (PP) defined as subjects in the ITT population taking study medication for 6 month and no identified as a major protocol violator.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 64 | 67
units on a scale
  Month 3 Mean Score | 0.78 (0.79) | 0.19 (0.78)
  Month 6 Mean Score | 0.88 (0.86) | -0.30 (0.85)

13. Secondary Outcome: Panel Assessment of Improvement Distribution From Screening
Description: as for outcome 11
Time Frame: Baseline to Month 3 and Baseline to Month 6
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Greatly decreased (Month 3) | 0 | 0
  Moderately decreased (Month 3) | 1 | 0
  Slightly decreased (Month 3) | 3 | 14
  No change (Month 3) | 28 | 29
  Slightly increased (Month 3) | 33 | 28
  Moderately increased (Month 3) | 8 | 4
  Greatly increased (Month 3) | 0 | 0
  Greatly decreased (Month 6) | 0 | 1
  Moderately decreased (Month 6) | 0 | 4
  Slightly decreased (Month 6) | 6 | 29
  No Change (Month 6) | 40 | 32
  Slightly increased (Month 6) | 20 | 8
  Moderately increased (Month 6) | 5 | 1
  Greatly increased (Month 6) | 2 | 0

14. Secondary Outcome: The Percentage Change From Baseline in Dihydrotestosterone (DHT) at Month 3, 6, and 10
Description: Mean percent change from Baseline for DHT. DHT was measured in pg/ml. Change from baseline = Month 3, 6, and 10 values minus baseline value.
Time Frame: Month 3, Month 6 and Month 10
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Percent change
  % Change in DHT - Month 3 | -16.92 (54.14) | -1.90 (47.58)
  % Change in DHT - Month 6 | -4.30 (38.73) | 22.83 (45.30)
  % Change in DHT - Month 10 | 3.85 (44.34) | 7.58 (50.28)

15. Secondary Outcome: The Percentage Change From Baseline in Testosterone at Month 3, 6, and 10
Description: Mean percent change from Baseline for testosterone. Testosterone was measured in ng/ml.
Time Frame: Month 3, Month 6, and Month 10
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Percent change
  % Change in Testosterone - Month 3 | 18.78 (28.69) | -5.27 (28.90)
  % Change in Testosterone - Month 6 | 8.15 (30.18) | -6.59 (31.86)
  % Change in Testosterone - Month 10 | 12.18 (26.17) | 0.99 (27.42)

16. Secondary Outcome: Endocrinology Shifts in Thyroid Stimulating Hormone (TSH), Thyroxine (T4), Prostate Specific Antigen (PSA), DHT, Testosterone (T), and Luteinizing Hormone (LH) From Baseline to Month 6 and Month 10.
Description: Normal ranges: TSH, 0.25-3.50 µIU/mL; T4, 4.5-12.0 mg/dL; PSA, ≤4 ng/mL; DHT, males (m): prepuberty, <0.1, adult, 0.25-0.75; females (f): prepuberty, <0.03, premenopausal, 0.05-0.3, menopausal, <0.03 ng/mL; T, m: 2.36-9.96; f: 0.08-0.86 ng/mL; LH, m: 1-8; f: follicular, 4-12; periovulatory, >20; luteal 5-20; postmenopausal, >10 IU/L.
Time Frame: Baseline to Month 6 and Month 10
Population: Intent to Treat (ITT) population defined as all randomized subjects received at least one dose of study mediction and having at least one on visit endpoint. LH was only assessed at baseline.
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  TSH - Baseline - Normal | 70 | 75
  TSH - Baseline - Abnormal | 3 | 0
  TSH - Month 6 - Normal | 70 | 69
  TSH - Month 6 - Abnormal | 0 | 4
  TSH - Month 10 - Normal | 71 | 74
  TSH - Month 10 - Abnormal | 1 | 1
  T4 - Baseline - Normal | 73 | 75
  T4 - Baseline - Abnormal | 0 | 0
  T4 - Month 6 - Normal | 70 | 71
  T4 - Month 6 - Abnormal | 0 | 2
  T4 - Month 10 - Normal | 72 | 74
  T4 - Month 10 - Abnormal | 0 | 1
  PSA - Screening - Normal | 73 | 75
  PSA - Screening - Abnormal | 0 | 0
  PSA - Month 6 - Normal | 70 | 73
  PSA - Month 6 - Abnormal | 0 | 0
  PSA - Month 10 - Normal | 72 | 75
  PSA - Month 10 - Abnormal | 0 | 0
  DHT - Screening - Normal | 72 | 74
  DHT - Screening - Abnormal | 1 | 1
  DHT - Month 6 - Normal | 69 | 69
  DHT - Month 6 - Abnormal | 1 | 4
  DHT - Month 10 - Normal | 70 | 72
  DHT - Month 10 - Abnormal | 2 | 3
  Testosterone - Screening - Normal | 73 | 74
  Testosterone - Screening - Abnormal | 0 | 1
  Testosterone - Month 6 - Normal | 67 | 71
  Testosterone - Month 6 - Abnormal | 3 | 2
  Testosterone - Month 10 - Normal | 69 | 74
  Testosterone - Month 10 - Abnormal | 3 | 1
  LH - Baseline - Normal | 67 | 64
  LH - Baseline - Abnormal | 6 | 11

17. Secondary Outcome: Laboratory Values: Electrolytes Assessed at Baseline and 6 Months.
Description: Sodium, Potassium (mEq/L), and Bicarbonate
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
mmol/L
  Sodium - Baseline | 141.23 (1.72) | 141.41 (1.62)
  Sodium - Month 6 | 141.54 (2.01) | 141.58 (1.65)
  Potassium (mEq/L) - Baseline | 4.22 (0.31) | 4.34 (0.33)
  Potassium (mEq/L) - Month 6 | 4.25 (0.32) | 4.29 (0.26)
  Bicarbonate - Baseline | 27.66 (2.19) | 28.23 (2.28)
  Bicarbonate - Month 6 | 26.61 (2.12) | 27.08 (2.30)

18. Secondary Outcome: Laboratory Values: Hematology Assessed at Baseline and 6 Months.
Description: Comparing Lab values and differences from Baseline to month 6
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: thousands/microliter
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
thousands/microliter
  WBC - Baseline | 6898.49 (1991.34) | 6336.93 (1815.00)
  WBC - Month 6 | 6463.61 (1421.58) | 6387.03 (1828.81)
  Neutrophils - Baseline | 53.46 (9.17) | 53.52 (8.63)
  Neutrophils - Month 6 | 52.47 (8.46) | 52.90 (8.51)
  Lymphocytes - Baseline | 35.96 (8.03) | 35.87 (8.28)
  Lymphocytes - Month 6 | 36.96 (7.61) | 36.03 (8.19)
  Monocytes - Baseline | 7.03 (1.64) | 7.03 (1.80)
  Monocytes - Month 6 | 7.08 (1.39) | 7.14 (1.75)
  Eosinophils - Baseline | 2.81 (2.34) | 2.69 (1.71)
  Eosinophils - Month 6 | 2.75 (2.08) | 2.99 (2.21)
  Basophils - Baseline | 0.48 (0.28) | 0.52 (0.28)
  Basophils - Month 6 | 0.50 (0.21) | 0.51 (0.26)
  Platelets - Baseline | 249.63 (52.79) | 250.19 (53.67)
  Platelets - Month 6 | 243.69 (46.03) | 240.26 (50.90)
  Hemoglobin (%)- Baseline | 15.44 (1.17) | 15.54 (0.88)
  Hemoglobin (%) - Month 6 | 15.41 (1.10) | 15.46 (0.86)
  MCV (fL)- Baseline | 92.12 (3.31) | 91.89 (4.06)
  MCV (fL) - Month 6 | 91.57 (3.51) | 91.44 (3.88)

19. Secondary Outcome: Laboratory Values: Liver Enzymes Assessed at Baseline and 6 Months.
Description: sGOT (AST)- serum Glutamic-Oxaloacetic Transaminase, sGPT (ALT) - serum Glutamic-Pyruvic Transaminase, Alkaline Phosphatase, Bilirubin(mg/dL) and Albumin(g/dL)
Time Frame: Baseline and Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
IU/L
  AST(SGOT) - Baseline | 23.10 (6.77) | 22.80 (6.14)
  AST(SGOT) - Month 6 | 25.88 (10.55) | 25.11 (9.51)
  ALT(SGPT) - Baseline | 29.79 (15.11) | 26.91 (12.36)
  ALT(SGPT) - Month 6 | 34.00 (25.79) | 30.47 (18.81)
  Alkaline Phosphatase - Baseline | 87.34 (40.14) | 85.79 (46.15)
  Alkaline Phosphatase - Month 6 | 85.51 (33.09) | 84.24 (42.44)
  Bilirubin (mg/dL) - Baseline | 0.78 (0.32) | 0.71 (0.28)
  Bilirubin (mg/dL) - Month 6 | 0.80 (0.32) | 0.79 (0.31)
  Albumin (g/dL) - Baseline | 4.66 (0.22) | 4.60 (0.25)
  Albumin (g/dL) - Month 6 | 4.64 (0.21) | 4.60 (0.24)

20. Secondary Outcome: Laboratory Values: Other Chemistry Assessed at Baseline and 6 Months.
Description: Glucose, Creatinine, Ferritine (ug/L) and Zinc (Hmol/L)
Time Frame: Baseline and Month 6
Population: Intent to Treat(ITT) population defined as all randomized subjects received at least one dose of study medication and having at least one on visit endpoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
mg/dL
  Glucose - Baseline | 104.48 (25.32) | 101.56 (16.17)
  Glucose - Month 6 | 104.49 (24.45) | 106.31 (20.82)
  Creatinine - Baseline | 1.03 (0.14) | 1.03 (0.14)
  Creatinine - Month 6 | 1.05 (0.11) | 1.06 (0.14)
  Ferritine (ug/L) - Baseline | 100.21 (55.11) | 131.91 (77.74)
  Ferritine (ug/L) - Month 6 | 109.61 (64.29) | 132.36 (87.91)
  Zinc (Hmol/L) - Baseline | 111.19 (35.35) | 112.66 (45.62)
  Zinc (Hmol/L) - Month 6 | 118.07 (40.75) | 113.87 (39.80)

21. Secondary Outcome: Sexual Function Inventory - Screening - Sex Drive, Erection, and Ejaculation
Description: In the past 7 days, to what extent have you considered: a lack of sex drive to be a problem?, your ability to get and keep erections to be a problem? your ejaculation to be a problem?
Time Frame: Screening
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Sex Drive - No Problem | 60 | 58
  Sex Drive - Very Small Problem | 5 | 5
  Sex Drive - Small Problem | 4 | 9
  Sex Drive - Medium Problem | 4 | 3
  Sex Drive - Big Problem | 0 | 0
  Erection - No Problem | 62 | 60
  Erection - Very Small Problem | 7 | 6
  Erection - Small Problem | 4 | 7
  Erection - Medium Problem | 0 | 2
  Erection - Big Problem | 0 | 0
  Ejaculation - No Problem | 64 | 63
  Ejaculation - Very Small Problem | 6 | 4
  Ejaculation - Small Problem | 3 | 7
  Ejaculation - Medium Problem | 0 | 1
  Ejaculation - Big Problem | 0 | 0

22. Secondary Outcome: Sexual Function Inventory - Baseline - Sex Drive, Erection, and Ejaculation
Description: as for outcome 21
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Sex Drive - No Problem | 63 | 60
  Sex Drive - Very small problem | 4 | 5
  Sex Drive - Small problem | 6 | 8
  Sex Drive - Medium problem | 0 | 1
  Sex Drive - Big problem | 0 | 0
  Erection - No Problem | 64 | 60
  Erection - Very small problem | 5 | 6
  Erection - Small problem | 4 | 7
  Erection - Medium problem | 0 | 1
  Erection - Big problem | 0 | 0
  Ejaculation - No Problem | 63 | 62
  Ejaculation - Very small problem | 7 | 5
  Ejaculation - Small problem | 3 | 7
  Ejaculation - Medium problem | 0 | 0
  Ejaculation - Big problem | 0 | 0

23. Secondary Outcome: Sexual Function Inventory - Month 3 - Sex Drive, Erection, and Ejaculation
Description: as for outcome 21
Time Frame: Month 3
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Sex Drive - No Problem | 49 | 59
  Sex Drive - Very small Problem | 12 | 8
  Sex Drive - Small Problem | 5 | 5
  Sex Drive - Medium Problem | 5 | 0
  Sex Drive - Big Problem | 0 | 1
  Erection - No Problem | 52 | 56
  Erection - Very Small Problem | 11 | 10
  Erection - Small Problem | 2 | 3
  Erection - Medium Problem | 6 | 3
  Erection - Big Problem | 0 | 1
  Ejaculation - No Problem | 55 | 59
  Ejaculation - Very Small Problem | 9 | 8
  Ejaculation - Small Problem | 3 | 3
  Ejaculation - Medium Problem | 4 | 2
  Ejaculation - Big Problem | 0 | 1

24. Secondary Outcome: Sexual Function Inventory - Month 6 - Sex Drive, Erection, and Ejaculation
Description: as for outcome 21
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Sex Drive - No Problem | 56 | 59
  Sex Drive - Very Small Problem | 7 | 6
  Sex Drive - Small Problem | 7 | 8
  Sex Drive - Medium Problem | 2 | 2
  Sex Drive - Big Problem | 0 | 0
  Erection - No Problem | 57 | 58
  Erection - Very Small Problem | 6 | 9
  Erection - Small Problem | 6 | 7
  Erection - Medium Problem | 3 | 1
  Erection - Big Problem | 0 | 0
  Ejaculation - No Problem | 58 | 59
  Ejaculation - Very Small Problem | 8 | 8
  Ejaculation - Small Problem | 4 | 6
  Ejaculation - Medium Problem | 2 | 2
  Ejaculation - Big Problem | 0 | 0

25. Secondary Outcome: Sexual Function Inventory - Month 10 - Sex Drive, Erection, and Ejaculation
Description: as for outcome 21
Time Frame: Month 10
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  Sex Drive - No Problem | 62 | 62
  Sex Drive - Very Small Problem | 7 | 6
  Sex Drive - Small Problem | 2 | 4
  Sex Drive - Medium Problem | 1 | 3
  Sex Drive - Big Problem | 0 | 0
  Erection - No Problem | 59 | 60
  Erection - Very Small Problem | 9 | 11
  Erection - Small Problem | 4 | 2
  Erection - Medium Problem | 0 | 2
  Erection - Big Problem | 0 | 0
  Ejaculation - No Problem | 60 | 62
  Ejaculation - Very Small Problem | 7 | 10
  Ejaculation - Small Problem | 4 | 1
  Ejaculation - Medium Problem | 0 | 2
  Ejaculation - Big Problem | 1 | 0

26. Secondary Outcome: Sexual Function Inventory: Shifts From Baseline to Month 6 in Sex Drive
Description: In the past 7 days, to what extent have you considered: a lack of sex drive to be a problem?, your ability to get and keep erections to be a problem? your ejaculation to be a problem? For example, "No Problem shift to No Problem" indicates that the participant experienced no problem at baseline and no problem at Month 6, respectively.
Time Frame: Baseline to Month 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No Problem shift to No Problem | 53 | 52
  No Problem shift to Very Small Problem | 6 | 4
  No Problem shift to Small Problem | 2 | 4
  No Problem shift to Medium Problem | 1 | 0
  No Problem shift to Big Problem | 0 | 0
  Very Small Problem shift to No Problem | 0 | 4
  Very Small Problem shift to Very Small Problem | 0 | 0
  Very Small Problem shift to Small Problem | 3 | 1
  Very Small Problem shift to Medium Problem | 1 | 0
  Very Small Problem shift to Big Problem | 0 | 0
  Small Problem shift to No Problem | 3 | 1
  Small Problem shift to Very Small Problem | 1 | 2
  Small Problem shift to Small Problem | 2 | 3
  Small Problem shift to Medium Problem | 0 | 2
  Small Problem shift to Big Problem | 0 | 0
  Medium Problem shift to No Problem | 0 | 1
  Medium Problem shift to Very Small Problem | 0 | 0
  Medium Problem shift to Small Problem | 0 | 0
  Medium Problem shift to Medium Problem | 0 | 0
  Medium Problem shift to Big Problem | 0 | 0
  Big Problem shift to No Problem | 0 | 0
  Big Problem shift to Very Small Problem | 0 | 0
  Big Problem shift to Small Problem | 0 | 0
  Big Problem shift to Medium Problem | 0 | 0
  Big Problem shift to Big Problem | 0 | 0

27. Secondary Outcome: Sexual Function Inventory: Shifts From Baseline to Month 6 - Erection
Description: as for outcome 26
Time Frame: Baseline to Month 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No Problem shift to No Problem | 53 | 52
  No Problem shift to Very Small Problem | 6 | 5
  No Problem shift to Small Problem | 3 | 3
  No Problem shift to Medium Problem | 1 | 0
  No Problem shift to Big Problem | 0 | 0
  Very Small Problem shift to No Problem | 2 | 3
  Very Small Problem shift to Very Small Problem | 0 | 3
  Very Small Problem shift to Small Problem | 2 | 0
  Very Small Problem shift to Medium Problem | 1 | 0
  Very Small Problem shift to Big Problem | 0 | 0
  Small Problem shift to No Problem | 2 | 1
  Small Problem shift to Very Small Problem | 0 | 1
  Small Problem shift to Small Problem | 1 | 4
  Small Problem shift to Medium Problem | 1 | 1
  Small Problem shift to Big Problem | 0 | 0
  Medium Problem shift to No Problem | 0 | 1
  Medium Problem shift to Very Small Problem | 0 | 0
  Medium Problem shift to Small Problem | 0 | 0
  Medium Problem shift to Medium Problem | 0 | 0
  Medium Problem shift to Big Problem | 0 | 0
  Big Problem shift to No Problem | 0 | 0
  Big Problem shift to Very Small Problem | 0 | 0
  Big Problem shift to Small Problem | 0 | 0
  Big Problem shift to Medium Problem | 0 | 0
  Big Problem shift to Big Problem | 0 | 0

28. Secondary Outcome: Sexual Function Inventory: Shifts From Baseline to Month 6 - Ejaculation
Description: as for outcome 26
Time Frame: Baseline to Month 6
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No Problem shift to No Problem | 54 | 54
  No Problem shift to Very Small Problem | 5 | 5
  No Problem shift to Small Problem | 2 | 3
  No Problem shift to Medium Problem | 1 | 0
  No Problem shift to Big Problem | 0 | 0
  Very Small Problem shift to No Problem | 3 | 3
  Very Small Problem shift to Very Small Problem | 3 | 1
  Very Small Problem shift to Small Problem | 1 | 0
  Very Small Problem shift to Medium Problem | 0 | 1
  Very Small Problem shift to Big Problem | 0 | 0
  Small Problem shift to No Problem | 1 | 1
  Small Problem shift to Very Small Problem | 0 | 2
  Small Problem shift to Small Problem | 1 | 3
  Small Problem shift to Medium Problem | 1 | 1
  Small Problem shift to Big Problem | 0 | 0
  Medium Problem shift to No Problem | 0 | 0
  Medium Problem shift to Very Small Problem | 0 | 0
  Medium Problem shift to Small Problem | 0 | 0
  Medium Problem shift to Medium Problem | 0 | 0
  Medium Problem shift to Big Problem | 0 | 0
  Big Problem shift to No Problem | 0 | 0
  Big Problem shift to Very Small Problem | 0 | 0
  Big Problem shift to Small Problem | 0 | 0
  Big Problem shift to Medium Problem | 0 | 0
  Big Problem shift to Big Problem | 0 | 0

29. Secondary Outcome: Sexual Function Inventory: Shifts From Baseline to Month 10 in Sex Drive
Description: as for outcome 26
Time Frame: Baseline to Month 10
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No Problem shift to No Problem | 57 | 55
  No Problem shift to Very Small Problem | 5 | 3
  No Problem shift to Small Problem | 0 | 0
  No Problem shift to Medium Problem | 0 | 2
  No Problem shift to Big Problem | 0 | 0
  Very Small Problem shift to No Problem | 2 | 4
  Very Small Problem shift to Very Small Problem | 1 | 0
  Very Small Problem shift to Small Problem | 1 | 1
  Very Small Problem shift to Medium Problem | 0 | 0
  Very Small Problem shift to Big Problem | 0 | 0
  Small Problem shift to No Problem | 3 | 1
  Small Problem shift to Very Small Problem | 1 | 3
  Small Problem shift to Small Problem | 1 | 3
  Small Problem shift to Medium Problem | 1 | 1
  Small Problem shift to Big Problem | 0 | 0
  Medium Problem shift to No Problem | 0 | 1
  Medium Problem shift to Very Small Problem | 0 | 0
  Medium Problem shift to Small Problem | 0 | 0
  Medium Problem shift to Medium Problem | 0 | 0
  Medium Problem shift to Big Problem | 0 | 0
  Big Problem shift to No Problem | 0 | 0
  Big Problem shift to Very Small Problem | 0 | 0
  Big Problem shift to Small Problem | 0 | 0
  Big Problem shift to Medium Problem | 0 | 0
  Big Problem shift to Big Problem | 0 | 0

30. Secondary Outcome: Sexual Function Inventory: Shifts From Baseline to Month 10 - Erection
Description: as for outcome 26
Time Frame: Baseline to Month 10
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No Problem shift to No Problem | 54 | 54
  No Problem shift to Very Small Problem | 6 | 5
  No Problem shift to Small Problem | 3 | 0
  No Problem shift to Medium Problem | 0 | 1
  No Problem shift to Big Problem | 0 | 0
  Very Small Problem shift to No Problem | 2 | 2
  Very Small Problem shift to Very Small Problem | 3 | 4
  Very Small Problem shift to Small Problem | 0 | 0
  Very Small Problem shift to Medium Problem | 0 | 0
  Very Small Problem shift to Big Problem | 0 | 0
  Small Problem shift to No Problem | 3 | 2
  Small Problem shift to Very Small Problem | 0 | 2
  Small Problem shift to Small Problem | 1 | 2
  Small Problem shift to Medium Problem | 0 | 1
  Small Problem shift to Big Problem | 0 | 0
  Medium Problem shift to No Problem | 0 | 1
  Medium Problem shift to Very Small Problem | 0 | 0
  Medium Problem shift to Small Problem | 0 | 0
  Medium Problem shift to Medium Problem | 0 | 0
  Medium Problem shift to Big Problem | 0 | 0
  Big Problem shift to No Problem | 0 | 0
  Big Problem shift to Very Small Problem | 0 | 0
  Big Problem shift to Small Problem | 0 | 0
  Big Problem shift to Medium Problem | 0 | 0
  Big Problem shift to Big Problem | 0 | 0

31. Secondary Outcome: Sexual Function Inventory: Shifts From Baseline to Month 10 - Ejaculation
Description: as for outcome 26
Time Frame: Baseline to Month 10
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dutasteride | Placebo
Number analyzed (Participants) | 73 | 75
Participants
  No Problem shift to No Problem | 56 | 56
  No Problem shift to Very Small problem | 2 | 6
  No Problem shift to Small Problem | 3 | 0
  No Problem shift to Medium Problem | 0 | 0
  No Problem shift to Big Problem | 1 | 0
  Very Small Problem shift to No Problem | 2 | 3
  Very Small Problem shift to Very Small Problem | 5 | 1
  Very Small Problem shift to Small Problem | 0 | 0
  Very Small Problem shift to Medium Problem | 0 | 1
  Very Small Problem shift to Big Problem | 0 | 0
  Small Problem shift to No Problem | 2 | 2
  Small Problem shift to Very Small Problem | 0 | 3
  Small Problem shift to Small Problem | 1 | 1
  Small Problem shift to Medium Problem | 0 | 1
  Small Problem shift to Big Problem | 0 | 0
  Medium Problem shift to No Problem | 0 | 0
  Medium Problem shift to Very Small Problem | 0 | 0
  Medium Problem shift to Small Problem | 0 | 0
  Medium Problem shift to Medium Problem | 0 | 0
  Medium Problem shift to Big Problem | 0 | 0
  Big Problem shift to No Proble | 0 | 0
  Big Problem shift to Very Small Problem | 0 | 0
  Big Problem shift to Small Problem | 0 | 0
  Big Problem shift to Medium Problem | 0 | 0
  Big Problem shift to Big Problem | 0 | 0

ADVERSE EVENTS:
Arm/Group | Dutasteride | Placebo
Serious Adverse Events (participants affected / at risk) | 0 | 1
Other Adverse Events (participants affected / at risk) | 12/73 | 7/75
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Dutasteride | Placebo
Thyroid Cancer (Endocrine disorders) | 0/73 (0) | 1/75 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dutasteride (N=73) | Placebo (N=75)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 12 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will no prohibit any investigator form publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.